CLINICAL TRIAL: NCT01744028
Title: A 52-week Multi-center Randomized Trial to Evaluate Remote Patient Monitoring Using the EXACT Patient-reported Outcome Tool on Reduction of Hospitalizations From Exacerbations in Patients With Chronic Obstructive Pulmonary Disease as Compared to Those Managed by Usual Care
Brief Title: Compare the Effect of a Remote Monitoring System Using the EXACT Tool to Reduce Hospitalizations Due to Chronic Obstructive Pulmonary Disease (COPD) Exacerbations. EXACT = Exacerbations of Chronic Pulmonary Disease Tool.
Acronym: PREMIERE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CIDD001D2401
Record Dates: First submitted 2012-12-04; First posted 2012-12-06 (Estimated); Last update posted 2020-12-10 (Actual); Status verified 2014-02

CONDITIONS: Remote Patient Monitoring in COPD Patients
Keywords: COPD, remote patient monitoring, Hub, exacerbations, EXACT
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Remote patient monitoring (Experimental): Remote patient monitoring system including the Exacerbations of Chronic Pulmonary Disease Tool (EXACT) tool can use changes in daily scores over a certain threshold level to alert notification to the clinical site. The site will contact the patient in order to determine the clinical significance associated with the change in score, and to treat the patient based on clinical judgment and clinical practice.
  Interventions: Device: Remote Patient Monitoring
- Usual care (Experimental): This group of patient will continue on their usual standard care as close to real life situation as possible.
  Interventions: Other: Usual care

INTERVENTIONS:
Device: Remote Patient Monitoring — Remote patient monitoring system including exacerbations of chronic pulmonary disease Tool - Patient Reported Outcome (EXACT PRO), Lung Monitor, and Pulse Oximeter
  Arms: Remote patient monitoring
Other: Usual care — Patients in the usual care arm will continue their normally established procedures of nurse/physician contact and evaluation, as is considered standard for each individual practitioner in the study.
  Arms: Usual care

SUMMARY:
The purpose of this pilot study is to evaluate a remote patient monitoring (RPM) system using a daily PRO tool (EXACT = Exacerbations of Chronic Pulmonary Disease Tool), in preventing hospitalization from Chronic Obstructive Pulmonary Disease (COPD) exacerbations in a COPD population at high risk of exacerbation, compared to those managed by usual care.

DETAILED DESCRIPTION:
This study uses two parallel groups of approximately 100 patients in each arm. After a screening period to confirm eligibility, patients will be randomized to either the RPM system group, or the usual care group. Both groups will be followed for 52 weeks until the end of study. There are only 4 planned study visits and patients will continue on their usual treatment.

The remote patient monitoring system will issue an alert to the clinical site once the established threshold change has been reached. The alert notification will require the clinical site to contact the patient and treat the patient based on clinical judgment and clinical practice. Patients in the usual care arm will be managed through their normally nurse/physician contact.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients with a diagnosis of Chronic Obstructive Pulmonary Disease (COPD), GOLD grade 2 or higher as classified by the Global Initiative for Chronic Obstructive Lung Disease (GOLD) guidelines, Updated 2011, including:
* Current or ex-smokers with a smoking history of at least 10 pack years nt
* Post-bronchodilator Forced Expiratory Volume in one second (FEV1) < 80% of the predicted normal value within 12 months prior to screening or at screening
* Post-bronchodilator FEV1/FVC (Forced Vital Capacity) < 70% within 12 months prior to screening or at screening
* A documented history of at least 2 COPD exacerbations requiring treatment with systemic corticosteroids and/or antibiotics in the previous 12 months prior to the screening visit, at least one of which required hospitalization.

Exclusion criteria:

* Use of investigational drugs at the time of enrollment, or within 30 days or 5 half-lives of enrollment, whichever is longer.
* Patients who have a COPD exacerbation not clinically resolved within 30 days prior to screening.
* Patients with a history of asthma, indicated by (but not limited to) the onset of respiratory symptoms suggestive of asthma (such as cough, wheezing, shortness of breath) prior to age 40 years.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2012-06; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
The number of hospitalizations and emergency room visits for management of COPD exacerbation(s) | 52 weeks
  Comparison of the total number of hospitalizations and emergency room visits (combined) for management of Chronic Obstructive Pulmonary Disease (COPD) exacerbation(s) between the two arms

SECONDARY OUTCOMES:
Lenght of hospitalization | 52 weeks
  Comparison of the average length of hospital stay for management of COPD exacerbation(s) between the two arms.
Time to first hospitalization | 52 weeks
  Comparison of the time to first occurrence of hospitalization for management of COPD exacerbation(s) between the two arms.
Use of health care resources | 52 weeks
  Comparison of the combined health care resource utilization (hospitalizations, unscheduled, scheduled office visits, telephone call contacts) for management of COPD between the two arms.
Number of medical visits | 52 weeks
  Comparison of the number of medical visits combined (hospitalizations, emergency room visits, unscheduled and scheduled office visits) for management of COPD between the two arms.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (16):
- Spain (10):
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Girona, Catalonia
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Catalonia
  - Novartis Investigative Site, Lleida, Catalonia
  - Novartis Investigative Site, Sant Boi de Llobregat, Catalonia
  - Novartis Investigative Site, Sant Cugat del Vallès, Catalonia
  - Novartis Investigative Site, Sant Joan Despí, Catalonia
  - Novartis Investigative Site, Majadanonda, Madrid
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Torremolinos
- Sweden (6):
  - Novartis Investigative Site, Gagnef
  - Novartis Investigative Site, Gothenburg
  - Novartis Investigative Site, Kungshamn
  - Novartis Investigative Site, Lund
  - Novartis Investigative Site, Östersund
  - Novartis Investigative Site, Stockholm

REFERENCES:
- See also: Results for CIDD001D2401 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=13123